CLINICAL TRIAL: NCT05835414
Title: Electroencephalogram (EEG) Enhanced Transcranial Magnetic Stimulation (eTMS) for Chronic Trauma and Stressor-Related Disorders (TSRD) (ETMS for Stress)
Brief Title: Electroencephalogram (EEG) Enhanced Transcranial Magnetic Stimulation (eTMS) for Chronic Trauma and Stressor-Related Disorders (TSRD)
Acronym: ETMS4Stress
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marcia Bockbrader, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Marcia Bockbrader, MD PhD, Principal Investigator, BEP Medical Group, LLC
Organization: BEP Medical Group, LLC (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEP-001
Expanded Access: Available
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Trauma and Stressor Related Disorders
Keywords: Transcranial Magnetic Stimulation; Chronic Trauma and Stressor Related Disorders; Veterans RAND 36-item health survey (VR-36); Health Related Quality of Life; EEG; Alpha Rhythms
MeSH Terms: conditions — Trauma and Stressor Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This will be a staged, open-label, Phase II/III safety, feasibility, and efficacy investigational device trial. A staged approach will be utilized to assess safety, feasibility, and preliminary efficacy with 30 participants with an interim analysis after data collection at 6 weeks. If safety benchmarks are passed, the study will proceed with Stage 2, in which an additional 270 participants will be enrolled using randomization to multiple baselines for efficacy analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adjunctive eTMS treatment (no delay) (Experimental): 6 weeks (30 sessions) of daily eTMS as an adjunct to standard of care TSRD treatment
  Interventions: Device: Adjunctive, midline prefrontal, lower intensity, shorter session, EEG-enhanced, repetitive transcranial magnetic stimulation (eTMS)

INTERVENTIONS:
Device: Adjunctive, midline prefrontal, lower intensity, shorter session, EEG-enhanced, repetitive transcranial magnetic stimulation (eTMS) — Approximately 2000 pulses per session (x30 sessions) of midline prefrontal, repetitive transcranial magnetic stimulation at 50% or less of motor threshold, calibrated via EEG to a resonant alpha frequency of the participant, and given over approximately 12 minutes. Given as an adjunct to standard of care and integrative treatment for TSRD.

SUMMARY:
The goal of this clinical trial is to learn about the safety, feasibility, and preliminary efficacy of EEG-enhanced transcranial magnetic stimulation (eTMS) as an adjunct to standard-of-care therapies for chronic trauma and stressor related disorders (TSRD) among US military veterans.

The main questions the study aims to answer are:

* Is it safe to provide 30 sessions of eTMS for veterans with chronic TSRD?
* Is it feasible to provide 30 sessions of eTMS as an adjunct to standard-of-care therapies for veterans with chronic TSRD?
* Does health-related quality of life improve among veterans after 30 sessions of eTMS as an adjunct to standard-of-care therapies for chronic TSRD?

Participants will undergo 30 sessions of eTMS as an adjunct to standard-of-care therapies for veterans with chronic TSRD, weekly reassessment during treatment, and intermittent follow-up for 36 weeks post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Positive identification as a Veteran per discharge paperwork (DD-214, DD-215, NGB-22, NGB-22A) and photo ID, or Veterans Health Administration Veteran Health Identification Card (VHIC)
* Presence of deployment-related stressful events (as defined by the Deployment Risk & Resilience Inventory-2, DRRI-2)
* Trauma event(s) (defined on the Life Experiences Checklist for DSM-5, LEC-5)
* Presence of 6 months or more of 6 or more "moderate" or worse symptoms from any of the five categories associated with stress disorders as operationalized on the PTSD Checklist for DSM-5 (PCL-5; intrusion, altered mood and cognitions, dissociation, avoidance, and arousal).
* Informed consent for study participation, off label-eTMS, and data use
* Enrollment in addiction services, if meets standard addiction treatment criteria
* Enrollment in opioid reduction services, if dependent on opioids and morphine equivalent daily dose exceeds 50 mg (50 morphine equivalent daily dose, MEDD)
* Agreement to limit daily alcoholic beverage consumption to no more than 2 servings
* Signed pain contract, if MEDD >= 80, per State of Ohio prescribing guidelines

Exclusion Criteria:

* Uncontrolled medical, psychological or neurological conditions including, but not limited to:
* Uncontrolled psychosis or mania
* Uncontrolled seizure disorder or EEG abnormalities that indicate risk of seizure, i.e., epileptiform discharges during the EEG recording
* Uncontrolled cardiac, pulmonary, or endocrine disorder (e.g., diabetes)
* Acute pain or illness
* Active, untreated addiction to prescription drugs, alcohol or illicit substances (not including cannabis or derivatives, which are available in many states under medical prescription or for recreational use)
* Clinically significant medical condition or abnormality that in the Investigator's judgment might pose a potential safety risk to the subject or limit the interpretation of the trial results
* Pregnant, or female unwilling to use effective birth control during the course of the trial (unless cleared for participation by obstetrician/gynecologist)
* Absolute contraindications to TMS: Presence of aneurysm clips or coils, cochlear or ocular implant, cortical epidural stimulator, deep brain stimulator, pacemaker or defibrillator, retained intracranial metal foreign body (bullets, shrapnel - excluding titanium and oral implants), steel stents or shunts, active vagal nerve stimulator, ventriculoperitoneal (VP) shunt.
* Prior TMS treatment
* Unwilling or unable to adhere to the study treatment, data collection schedule, or study procedures

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with device-related serious adverse events | 6 weeks
  To address safety of the procedure, the study investigators will report number of participants (of 30 initial cohort) with expected, device-related serious adverse events (SAE's) or unexpected, device-related SAE's during treatment
Rate of participants completing 80% of scheduled visits | 6 weeks
  To assess feasibility of the procedure, the study investigators will report the rate of participants (for initial cohort of 30) completing >= 80% of the 30 scheduled eTMS sessions

SECONDARY OUTCOMES:
Mean change in Veterans RAND 36-item health survey (VR-36) mental component scores (MCS) | 6 weeks
  To assess efficacy of the procedure to improve health related quality of life, the study investigators will report the mean change from baseline to week 6 in mental component score (MCS) on Veterans RAND 36-item health survey (VR-36) for participants (in initial cohort of 30) who completed >=80% of eTMS sessions

CONTACTS AND LOCATIONS:
Locations (1):
- BEP Medical Group LLC, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT05835414/ICF_000.pdf